CLINICAL TRIAL: NCT02538315
Title: Using 3,4-dihydroxy-6-[18F]-Fluoro-l-phenylalanine ( [18F]FDOPA) PET/CT to Monitor the Effectiveness of Fetal Dopaminergic Grafts in Parkinson Disease Patients
Brief Title: Using [18F]FDOPA PET/CT to Monitor the Effectiveness of Fetal Dopaminergic Grafts in Parkinson Disease Patients
Status: Terminated | Type: Observational
Why Stopped: lack of patients due to COVID
Sponsor: University of Saskatchewan (Other)
Collaborators: University of Manitoba (Other)
Responsible Party: Principal Investigator, Rajan Rakheja, Principal Investigator, University of Saskatchewan
Other Study IDs: Bio 15-21
Record Dates: First submitted 2015-08-25; First posted 2015-09-02 (Estimated); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Parkinson's Disease
Keywords: [18F]FODPA, Parkinson's, PET/CT, Stem Cell transplantation
MeSH Terms: conditions — Parkinson Disease | interventions — fluorodopa F 18

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgery plus PET/CT imaging: Dopaminergic stem cell transplant and [18F]FDOPA PET/CT
  Interventions: Drug: [18F]FDOPA PET/CT

INTERVENTIONS:
Drug: [18F]FDOPA PET/CT — Implantation of fetal dopaminergic stem cell transplantation by neuro-surgeon followed by [18F]FDOPA PET/CT imaging
  Other Names: F-18 Fluorodopa

SUMMARY:
While positron emission tomography/computed tomography (PET/CT) can assist in the diagnosis of Parkinson disease (PD), it can also potentially help monitor treatment options for PD. One such experimental therapeutic option for PD is fetal dopaminergic transplantation trials. A potential goal of such novel therapies is to replace deficient dopaminergic neurons in PD. Researchers at the University of Saskatchewan have been at the frontier of these exciting treatment options. [18F]FDOPA PET/CT imaging has been successfully used by some authors to monitor engraftment and assess efficacy of fetal dopaminergic transplant . This study also aims to utilize [18F]FDOPA PET/CT imaging to potentially aid in detecting alterations in the dopaminergic pathway from these innovative surgical treatment options.

There are two main objectives of this study: 1) Evaluate the effectiveness of fetal dopaminergic grafts in patients with PD using FDOPA PET imaging pre and post-surgical implantation and a secondary longer term goal 2) Correlate the [18F]FDOPA PET/CT findings in early PD with post-mortem pathological analyses of PD

DETAILED DESCRIPTION:
Since the progression of PD is in most cases inexorable, there is an urgent need for curative or restorative treatments, especially for patients whose response to pharmaceutical treatment is marred by levodopa-evoked dyskinesias, or intolerable on-off fluctuations. This project focuses on the option of surgical implantation of embryonic dopamine neurons. Despite promising reports in some early case studies, this daring approach has not always shown consistent clinical outcomes. The factors responsible for this state of affairs remain uncertain, although some studies showed significantly better clinical outcome in younger PD patients (≤ 60 years) as compared to older patients (≥ 60 years). In a number of small clinical studies, researchers at the University of Saskactchewan have shown one of the most consistent improvements in clinical outcomes in fetal dopaminergic grafts, as has been confirmed in a recent review of the literature. Follow-up FDOPA-PET studies have linked enhanced tracer uptake in target regions to persistent improvements in unified parkison disease rating scale (UPDRS), and FDOPA-PET is informative about the relationship between targeting of specific striatal regions and the occurrence of dyskinesias.

Co-aaplicants of this research study have received approval and funding to undertake a new clinical trial of fetal dopaminergic neurons for the treatment of advanced and otherwise refractory PD. The main objective of the present study is to correlate the clinical outcomes of PD patients who undergo fetal dopamine neuron transplantation in the new study protocol with changes in FDOPA-PET/CT. Neurologists at the University of Saskachewan and the Royal University Hospital-Saskatoon have assembled an extensive database of PD patients which have been followed prospectively for as long as a decade. As noted above, the relationship between FDOPA-PET/CT and post-mortem findings is poorly documented in small patient samples, even though autopsy findings remain the gold standard for differential diagnosis of parkinsonian syndromes, as noted above. The established reputations of these neurologists in the PD community continues to be an important prerequisite for brain banking in Saskatchewan, and an important side objective of this project is to integrate molecular imaging with prospective post mortem analysis of extensively-documented PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease based on clinical diagnosis by Neuro-surgeon and/or Neurologist with specialty in Parkinson's disease
* Must be a resident of Canada
* Able to understand and provide written informed consent
* Referred by a treating physician
* Patients must be able to tolerate the physical/logistical requirements of a FDOPA-PET/CT scan, including withholding of medication, lying supine for up to 45 minutes, and intravenous cannulation for injection of the study drug
* 18 years and older, with clinical diagnosis of PD (presence of two out of following three symptoms: bradykinesia, rigidity and resting tremor) as per standard clinical practice

Exclusion Criteria:

* Medically unstable patients (e.g. acute cardiac or respiratory distress or hypotensive, etc.)
* Patients who exceed the safe weight limit of the PET/CT bed or who cannot fit through the PET/CT bore
* Patients who are claustrophobic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's patients screened by Dr. I. Mendez
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Differences (assessed by standard uptake values (SUV)) between pre and post-surgical nigrostriatal uptake of [18F]FDOPA | 1-2 years
  Change in the distribution of [18F]FDOPA from pre and post surgical brain scan. We are hoping to see an improvement in [18F]FDOPA in the nigrostriatal dopamine following fetal dopaminergic grafts transplant

CONTACTS AND LOCATIONS:
Overall Officials: Rajan Rakheja, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- University Of Saskatchewan, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Result] Eshuis SA, Jager PL, Maguire RP, Jonkman S, Dierckx RA, Leenders KL. Direct comparison of FP-CIT SPECT and F-DOPA PET in patients with Parkinson's disease and healthy controls. Eur J Nucl Med Mol Imaging. 2009 Mar;36(3):454-62. doi: 10.1007/s00259-008-0989-5. Epub 2008 Nov 27. PMID 19037637